CLINICAL TRIAL: NCT00017563
Title: Phase I/II Study of Neoadjuvant Weekly Docetaxel and Mitoxantrone Prior to Prostatectomy in Patients With High Risk Localized Prostate Cancer
Brief Title: Combination Chemotherapy Followed by Surgery in Treating Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tom Beer, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068719; OHSU-2794 (Other: OHSU IRB); OHSU-HOR-00037-L; NCI-G01-1962
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Results first posted 2011-08-31 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage II prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel, Mitoxantrone, Conventional Surgery (Experimental): Drug: Docetaxel-35 mg/m2 i.v. over 15 - 30 minutes will be administered immediately after the mitoxantrone on the same schedule.
  Drug: Mitoxantrone-Initial dose will be 2 mg/m2 weekly for 3 of every 4 weeks. The dose will then be escalated as described in the dose escalation section up to a maximum dose of 6 mg/m2 weekly for 3 of every 4 weeks.
  Procedure/Surgery: Conventional Surgery- Prostatectomy will be scheduled 2-4 weeks after the last dose of chemotherapy
  Interventions: Drug: docetaxel; Drug: mitoxantrone hydrochloride; Procedure: conventional surgery

INTERVENTIONS:
Drug: docetaxel — 35 mg/m2 i.v. over 15 - 30 minutes will be administered immediately after the mitoxantrone on the same schedule.
Drug: mitoxantrone hydrochloride — Initial dose will be 2 mg/m2 weekly for 3 of every 4 weeks. The dose will then be escalated as described in the dose escalation section up to a maximum dose of 6 mg/m2 weekly for 3 of every 4 weeks.
Procedure: conventional surgery — Prostatectomy will be scheduled 2 - 4 weeks after the last dose of chemotherapy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving chemotherapy before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy followed by surgery in treating patients who have localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 5-year freedom from prostate-specific antigen (PSA) recurrence in patients treated with this regimen.
* Define the maximum tolerated dose of neoadjuvant docetaxel and mitoxantrone followed by prostatectomy in patients with high-risk localized prostate cancer. (Phase I completed as of 2/15/02)
* Determine the toxicity of this regimen in these patients.
* Determine the PSA response rate and pathologic response rate in patients treated with this regimen.
* Determine the clinical response in patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.
* Determine the surgical margin status at time of prostatectomy in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of mitoxantrone. (Phase I completed as of 2/15/02)

Patients receive neoadjuvant docetaxel and mitoxantrone weekly on weeks 1-3. Treatment repeats once a week for a total of 4 courses.

Patients receive escalating doses of mitoxantrone until the maximum tolerated dose is determined. (Phase I completed as of 2/15/02)

Patients undergo prostatectomy 2-4 weeks after completion of neoadjuvant chemotherapy.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * High-risk, as defined by 1 of the following:

    * Stage T2b (palpable bilateral involvement) or surgically resectable T3
    * PSA 15 ng/mL or greater
    * Gleason grade greater than 4+3 (4+3, 4+4, or 5+any, but not 3+4)
* At least a 50% chance of prostate cancer recurrence within 5 years
* Planned prostatectomy as primary therapy
* No evidence of bone metastases by bone scan
* No evidence of lymph nodes greater than 2 cm on pelvic computed tomography (CT) scan (scan required only if PSA greater than 40 ng/mL)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Eastern Cooperative Oncology Group(ECOG) 0-2

Life expectancy:

* At least 10 years

Hematopoietic:

* White Blood Cell(WBC) at least 3,000/mm^3
* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Conjugated bilirubin no greater than upper limit of normal (ULN)
* Alkaline phosphatase no greater than 4 times ULN
* Alanine transaminase(ALT) no greater than 2 times ULN (1.5 times ULN if alkaline phosphatase greater than 2.5 times ULN)

Renal:

* Not specified

Cardiovascular:

* Ejection fraction greater than 50% by Multiple Gated Acquisition(MUGA)scan

Other:

* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No significant active medical illness that would preclude study therapy
* No peripheral neuropathy grade 2 or greater
* No hypersensitivity to drugs formulated with polysorbate-80
* No significant contraindications to corticosteroids

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior cytotoxic chemotherapy
* No other concurrent cytotoxic chemotherapy

Endocrine therapy:

* No prior or concurrent conventional hormonal therapy

Radiotherapy:

* No prior or concurrent radiotherapy (external beam or brachytherapy)

Surgery:

* See Disease Characteristics

Other:

* No prior or concurrent cryotherapy

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2000-09; Primary Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz M. Beer, MD, Study Chair — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel and Mitox: Drug: docetaxel
  35 mg/m2 i.v. over 15 - 30 minutes will be administered immediately after the mitoxantrone on the same schedule.
  Drug: mitoxantrone hydrochloride
  Initial dose will be 2 mg/m2 weekly for 3 of every 4 weeks. The dose will then be escalated as described in the dose escalation section up to a maximum dose of 6 mg/m2 weekly for 3 of every 4 weeks.
Period: Overall Study
Arm/Group | Docetaxel and Mitox
Started | 57
Completed | 56
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel and Mitox
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.56 (6.279)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 57
Region of Enrollment [Number; unit: participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 5-year Freedom From Prostate Specific Antigen (PSA) Recurrence.
Description: Number of participants that experienced 5-year freedom from Prostate Specific Antigen (PSA) recurrence (PSA > 0.4 ng/ml confirmed by a second PSA that is higher than the first by any amount (2)) in men with high risk localized prostate cancer treated with neoadjuvant docetaxel/mitoxantrone followed by surgery.
Time Frame: Every 3 months after surgery for up to 5 years.
Measure: Number; unit: participants
Arm/Group | Docetaxel and Mitox
Number analyzed (Participants) | 57
participants | 30

ADVERSE EVENTS:
Arm/Group | Docetaxel and Mitox
Serious Adverse Events (participants affected / at risk) | 43/57
Other Adverse Events (participants affected / at risk) | 57/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel and Mitox (N=57)
Neutropenia (Blood and lymphatic system disorders) | 18
Leukopenia (Blood and lymphatic system disorders) | 21
Abdominal Pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel and Mitox (N=57)
Hyperglycemia (Metabolism and nutrition disorders) | 11
Dermatology-Skin Toxicity (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 10
Anemia (Blood and lymphatic system disorders) | 3
Fatigue (General disorders) | 8
Hypophosphatemia (Blood and lymphatic system disorders) | 5
Hyperlacrimation (Eye disorders) | 4
Onycholysis (Skin and subcutaneous tissue disorders) | 17
Taste Disturbance (General disorders) | 4
Vision (Eye disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No